CLINICAL TRIAL: NCT05656638
Title: Treatment of Grammatical Time Marking in Post-Stroke Aphasia: a Study of French-Speaking Subjects With Chronic Fluent and Non-fluent Aphasia
Brief Title: Treatment of Grammatical Time Marking in Post-Stroke Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Neuchatel (Other)
Responsible Party: Principal Investigator, Marion Fossard, Professor, University of Neuchatel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Unine2022-01807
Record Dates: First submitted 2022-12-01; First posted 2022-12-19 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Brain Injury, Vascular; Aphasia; Stroke
MeSH Terms: conditions — Cerebrovascular Trauma; Aphasia; Stroke | interventions — Speech Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain-injured participants (Experimental): Participants with post-stroke fluent or non-fluent chronic aphasia
  Interventions: Behavioral: Speech and language therapy

INTERVENTIONS:
Behavioral: Speech and language therapy — The treatment focuses on grammatical time marking. The aim of the treatment is to train underlying grammatical time marking processes, which were identified as deficient during a preliminary evaluation. The intervention is composed of 4 steps inspired by models and hypotheses from the literature on the subject. Step 1: "temporal adverbial selection", subject must identify the tense encoded in sentences and select the correct adverbial among those proposed. Step 2: "selection of inflected verb forms", subject must identify the tense encoded in the sentence and select the correct verb form among those proposed. Step 3: "production of inflected verb forms", subject must identify the tense encoded in the sentence and produce inflected verbs. Step 4: "semantic narration", subject must describe scenes using verbs inflected according to the previously defined reference time.

SUMMARY:
The study aims to assess an individual or self-administered computer therapy's effectiveness in grammatical time marking. The main objective is to examine whether the therapy improves grammatical time marking of inflected verbs treated on the sessions. We also explore whether the observed progress can be transferred to untrained items, more ecological contexts and if is maintained two and four weeks after the end of treatment.

This therapy will be administered to six individuals with brain lesions after stroke. Four individuals will take part of the individual therapy and two individuals will take part of the self-administered computer therapy. The therapy will last one month, at the rate of three weekly sessions of approximately one hour.

ELIGIBILITY:
Inclusion Criteria:

* Have had an imaging-objectified stroke in adulthood that resulted in aphasia (fluent or non-fluent). The time between the stroke and participation in this study must be greater than 6 months.
* Be a native French speaker or have excellent mastery of French.
* Be between 18 and 75 years old.
* Present grammatical tense marking disorders objectified by language evaluation (deficit scores on the "Batterie d'Évaluation de la Production Syntaxique" (BEPS) verb flexion task, Monetta et al., 2018; and/or on the "Test d'expression morpho-syntaxique fine" (T.E.M.F.) active sentence production subtask, Bernaert-Paul and Simonin, 2011).

Exclusion Criteria:

* Present chronic symptoms of a substance use disorder as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria.
* Have significant uncorrected vision and/or hearing impairment.
* Have significant impairments in oral/written comprehension.
* Present apraxia of speech or a severe arthritic disorder
* Present hemineglect
* Present impaired judgment and discernment, objectified by a neuropsychological evaluation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Change from the score on an inflected verb production task after the end of the therapy: treated items | Baselines, middle of the treatment (after 2 weeks of treatment), post-treatment (24-48 hours after the last session of the therapy)
  The inflected verb production task evaluates subject's ability to produce an inflected verb form according to time context given by a short sentence. The score is obtained by adding the points (0 or 1) obtained for each item and is calculated per time reference.
  The task will be administered three times before the therapy (baselines), once in the middle of the therapy (after 2 weeks of treatment) and directly (24-48 hours) after the last session of the therapy (post-treatment) to analyze the change of performance.
Change from time accuracy on a semantic narration task after the end of the therapy: treated semantic narrations | Baselines, middle of the treatment (after 2 weeks of treatment), post-treatment (24-48 hours after the last session of the therapy)
  The semantic narration task evaluates subject's ability to produce inflected verb forms according to time context. Semantic narrations are based on imagined stories and according to a given temporal frame. This task includes 2 pictorial sequences per temporal reference. The accuracy of time marking in semantic narration task is calculated using ratios.
  The task will be administered three times before the therapy (baselines), once in the middle of the therapy (after 2 weeks of treatment) and directly (24-48 hours) after the last session of the therapy (post-treatment) to analyze the change of performance.
Change from the score on an inflected verb production task after the end of the therapy: untreated items | Baselines, middle of the treatment (after 2 weeks of treatment), post-treatment (24-48 hours after the last session of the therapy)
  The inflected verb production task evaluates subject's ability to produce an inflected verb form according to time context given by a short sentence. The score is obtained by adding the points (0 or 1) obtained for each item and is calculated per time reference.
  The task will be administered three times before the therapy (baselines), once in the middle of the therapy (after 2 weeks of treatment) and directly (24-48 hours) after the last session of the therapy (post-treatment) to analyze the change of performance.
Change from time accuracy on a semantic narration task after the end of the therapy: untreated semantic narrations | Baselines, middle of the treatment (after 2 weeks of treatment), post-treatment (24-48 hours after the last session of the therapy)
  The semantic narration task evaluates subject's ability to produce inflected verb forms according to time context. Semantic narrations are based on imagined stories and according to a given temporal frame. This task includes 2 pictorial sequences per temporal reference. The accuracy of time marking in semantic narration task is calculated using ratios.
  The task will be administered three times before the therapy (baselines), once in the middle of the therapy (after 2 weeks of treatment) and directly (24-48 hours) after the last session of the therapy (post-treatment) to analyze the change of performance.
Change from the score on an inflected verb production task 2 and 4 weeks after the end of the therapy: treated items | Post-treatment (24-48 hours after the last session of the therapy), 2-4 weeks follow-up
  The inflected verb production task evaluates subject's ability to produce an inflected verb form according to time context given by a short sentence. The score is obtained by adding the points (0 or 1) obtained for each item and is calculated per time reference.
  The task will be administered directly (24-48 hours) after the last session of the therapy (post-treatment) and 2-4 weeks after the treatment (follow-up) to analyze the maintenance of performance.
Change from the score on an inflected verb production task 2 and 4 weeks after the end of the therapy: untreated items | Post-treatment (24-48 hours after the last session of the therapy), 2-4 weeks follow-up
  The inflected verb production task evaluates subject's ability to produce an inflected verb form according to time context given by a short sentence. The score is obtained by adding the points (0 or 1) obtained for each item and is calculated per time reference.
  The task will be administered directly (24-48 hours) after the last session of the therapy (post-treatment) and 2-4 weeks after the treatment (follow-up) to analyze the maintenance of performance.
Change from time accuracy on a semantic narration task 2 and 4 weeks after the end of the therapy: treated semantic narrations | Post-treatment (24-48 hours after the last session of the therapy), 2-4 weeks follow-up
  The semantic narration task evaluates subject's ability to produce inflected verb forms according to time context. Semantic narrations are based on imagined stories and according to a given temporal frame. This task includes 2 pictorial sequences per temporal reference. The accuracy of time marking in the semantic narration task is calculated using ratios.
  The task will be administered directly (24-48 hours) after the last session of the therapy (post-treatment) and 2-4 weeks after the treatment (follow-up) to analyze the maintenance of performance.
Change from time accuracy on a semantic narration task 2 and 4 weeks after the end of the therapy: untreated semantic narrations | Post-treatment (24-48 hours after the last session of the therapy), 2-4 weeks follow-up
  The semantic narration task evaluates subject's ability to produce inflected verb forms according to time context. Semantic narrations are based on imagined stories and according to a given temporal frame. This task includes 2 pictorial sequences per temporal reference. The accuracy of time marking in the semantic narration task is calculated using ratios.
  The task will be administered directly (24-48 hours) after the last session of the therapy (post-treatment) and 2-4 weeks after the treatment (follow-up) to analyze the maintenance of performance.
Change from the score on an inflected verb production task 2 and 4 weeks after the end of the therapy: treated items | Baselines, 2-4 weeks follow-up
  The inflected verb production task evaluates subject's ability to produce an inflected verb form according to time context given by a short sentence. The score is obtained by adding the points (0 or 1) obtained for each item and is calculated per time reference.
  The task will be administered three times before the therapy (baselines) and 2-4 weeks after the treatment (follow-up) to analyze the long-term change of performance.
Change from the score on an inflected verb production task 2 and 4 weeks after the end of the therapy: untreated items | Baselines, 2-4 weeks follow-up
  The inflected verb production task evaluates subject's ability to produce an inflected verb form according to time context given by a short sentence. The score is obtained by adding the points (0 or 1) obtained for each item and is calculated per time reference.
  The task will be administered three times before the therapy (baselines) and 2-4 weeks after the treatment (follow-up) to analyze the long-term change of performance.
Change from time accuracy on a semantic narration task 2 and 4 weeks after the end of the therapy: treated semantic narrations | Baselines, 2-4 weeks follow-up
  The semantic narration task evaluates subject's ability to produce inflected verb forms according to time context. Semantic narrations are based on imagined stories and according to a given temporal frame. This task includes 2 pictorial sequences per temporal reference. The accuracy of time marking in the semantic narration task is calculated using ratios.
  The task will be administered three times before the therapy (baselines) and 2-4 weeks after the treatment (follow-up) to analyze the long-term change of performance.
Change from time accuracy on a semantic narration task 2 and 4 weeks after the end of the therapy: untreated semantic narrations | Baselines, 2-4 weeks follow-up
  The semantic narration task evaluates subject's ability to produce inflected verb forms according to time context. Semantic narrations are based on imagined stories and according to a given temporal frame. This task includes 2 pictorial sequences per temporal reference. The accuracy of time marking in the semantic narration task is calculated using ratios.
  The task will be administered three times before the therapy (baselines) and 2-4 weeks after the treatment (follow-up) to analyze the long-term change of performance.

SECONDARY OUTCOMES:
Change from time accuracy on an episodic/procedural narration task after the end of the therapy | Baselines, middle of the treatment (after 2 weeks of treatment), post-treatment (24-48 hours after the last session of the therapy)
  The episodic/procedural narration task evaluates subject's ability to produce inflected verb forms according to time context in a narrative situation. This task is administered in order to analyze the transfer of the gains of the therapy to a more ecological context (as it is free of verbal or pictorial support). The accuracy of time marking in the semantic narration task is calculated using ratios.
  The task will be administered three times before the therapy (baselines), once in the middle of the therapy (after 2 weeks of treatment) and directly (24-48 hours) after the last session of the therapy (post-treatment) to analyze the change of performance.
Change from time accuracy on an episodic/procedural narration task 2 and 4 weeks after the end of the therapy | Post-treatment (24-48 hours after the last session of the therapy), 2-4 weeks follow-up
  The episodic/procedural narration task evaluates subject's ability to produce inflected verb forms according to time context in a narrative situation. This task is administered in order to analyze the transfer of the gains of the therapy to a more ecological context (as it is free of verbal or pictorial support). The accuracy of time marking in the semantic narration task is calculated using ratios.
  The task will be administered directly (24-48 hours) after the last session of the therapy (post-treatment) and 2-4 weeks after the treatment (follow-up) to analyze the maintenance of performance.
Change from time accuracy on an episodic/procedural narration task 2 and 4 weeks after the end of the therapy | Baselines, 2-4 weeks follow-up
  The episodic/procedural narration task evaluates subject's ability to produce inflected verb forms according to time context in a narrative situation. This task is administered in order to analyze the transfer of the gains of the therapy to a more ecological context (as it is free of verbal or pictorial support). The accuracy of time marking in the semantic narration task is calculated using ratios.
  The task will be administered three times before the therapy (baselines) and 2-4 weeks after the treatment (follow-up) to analyze the long-term change of performance.
Change at a control task after the end of the therapy | Baselines, middle of the treatment (after 2 weeks of treatment), post-treatment (24-48 hours after the last session of the therapy)
  The control task ensures that progress is specific to the treatment. This task is specific to each participant: it is a logopedic/neuropsychological test for which the participant has deficit scores and whose content is not influenced by the treatment (e.g., a test on calculation).
  The task will be administered three times before the therapy (baselines), once in the middle of the therapy (after 2 weeks of treatment) and directly (24-48 hours) after the last session of the therapy (post-treatment) to analyze the change of performance.
Change at a control task 2 and 4 weeks after the end of the therapy | Post-treatment (24-48 hours after the last session of the therapy), 2-4 weeks follow-up
  The control task ensures that progress is specific to the treatment. This task is specific to each participant: it is a logopedic/neuropsychological test for which the participant has deficit scores and whose content is not influenced by the treatment (e.g., a test on calculation).
  The task will be administered directly (24-48 hours) after the last session of the therapy (post-treatment) and 2-4 weeks after the treatment (follow-up) to analyze the maintenance of performance.
Change at a control task 2 and 4 weeks after the end of the therapy | Baselines, 2-4 weeks follow-up
  The control task ensures that progress is specific to the treatment. This task is specific to each participant: it is a logopedic/neuropsychological test for which the participant has deficit scores and whose content is not influenced by the treatment (e.g., a test on calculation).
  The task will be administered three times before the therapy (baselines) and 2-4 weeks after the treatment (follow-up) to analyze the long-term change of performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Neuchâtel, Neuchâtel, Switzerland